CLINICAL TRIAL: NCT03403114
Title: Vaccine Attitudes and Practices of Hospital Specialists
Acronym: SPECIVAC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Innovative clinical research network in vaccinology (I-REIVAC) (Unknown); Observatoire Régionale de la santé ORS-PACA (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI16019
Record Dates: First submitted 2017-12-11; First posted 2018-01-18 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Vaccine Practice
Keywords: Vaccine hesitancy; Hospital specialists (HS); Vaccination survey
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — a 15min questionnaire

SUMMARY:
This study aims to evaluate the perceptions and knowledge of hospital specialists regarding vaccine recommendations targeting their patients, to study their behavior with respect to these recommendations and to quantify their vaccine hesitancy.

ELIGIBILITY:
Inclusion Criteria:

* To be a physician in one of the participating institutions
* Or to be a contract physician in participating institutions

Exclusion Criteria:

* Interns
* Attached practitioners
* Emergency physicians

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Physicians with a frequent activity of practice and advice vaccines, called "vaccinators" (most medical specialties): 100% of those meeting the inclusion criteria will be contacted for inclusion
  * Physicians "no or weak vaccinators" (anesthesiologists, surgeons, psychiatrists…): 30% of those meeting the inclusion criteria will be chosen by drawing lots
Sampling Method: Non-Probability Sample
Enrollment: 1851 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Proportions of Hospital Specialists (HS) with knowledge of vaccine recommendations targeting their patients | 15 minutes
Proportions of HS regularly recommending recommended vaccines to their patients | 15 minutes
Proportions of HS with doubts about recommended vaccines | 15 minutes

SECONDARY OUTCOMES:
Link between perception of benefits and risks of vaccines, knowledge of vaccine-preventable diseases, trust in different sources of information and vaccine hesitancy will be measured by questionnaire (measure by multiple logistic regressions) | 15 minutes
Measure of attitudes and practices of HS vis-a-vis to vaccination and their specialty by questionnaire | 15 minutes
  number of HS vaccinator or not by specialty in connection with their attitudes and practices
Percentages of HS feeling sufficiently trained or confident to explain to patients about vaccines | 15 minutes
Percentages of HS claiming to be vaccinated, by type of vaccine | 15 minutes
Percentages of HS children reported vaccinated by type of vaccine | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, Professor, Principal Investigator — CIC 1417 Centre d'investigation clinique; Pierre VERGER, MD, Study Chair — ORS PACA UMR 912 SESSTIM
Locations (14):
- France (14):
  - CRC Annecy, Annecy
  - CIC Besançon, Besançon
  - CIC Clermont-Ferrand, Clermont-Ferrand
  - CIC Dijon, Dijon
  - CIC Lille, Lille
  - CIC Limoges, Limoges
  - Service d'Hygiène, Epidémiologie et Prévention, Groupement Hospitalier Edouard Herriot et Unité de recherche clinique ne Immunologie du centre hospitalier Lyon Sud, Lyon
  - CIC Montpellier, Montpellier
  - Service de maladies infectieuses Nancy, Nancy
  - Service de maladies infectieuses Nîmes, Nîmes
  - CIC Rennes, Rennes
  - CIC Strasbourg, Strasbourg
  - CIC Cochin Pasteur, Paris, Île-de-France Region
  - CIC Bichat, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No